CLINICAL TRIAL: NCT05893732
Title: Efficacy of High-Intensity Laser Therapy in the Management of Meralgia Paresthetica: a Randomized Controlled Trial
Brief Title: HILT for Meralgia Paresthetica
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy ElMeligie, Lecturer of Physical Therapy and Director of Electromyography Lab, Ahram Canadian University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 012/004277
Record Dates: First submitted 2023-05-30; First posted 2023-06-08 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Meralgia Paresthetica; Lateral Femoral Cutaneous Nerve Entrapment
MeSH Terms: conditions — Femoral Neuropathy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: In this study, both the participants and the outcomes assessor will be blinded. Participants will be unaware of whether they are receiving active HILT or sham HILT, while the outcomes assessor will not know the treatment allocation while assessing the outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-Intensity Laser Therapy (HILT) Group (Experimental): Participants in this group will receive High-Intensity Laser Therapy (HILT) treatment for Meralgia Paresthetica (MP).
  Interventions: Device: High-Intensity Laser Therapy (HILT)
- Sham High-Intensity Laser Therapy (Sham HILT) Group (Sham Comparator): Participants in this group will receive sham High-Intensity Laser Therapy (sham HILT) treatment for Meralgia Paresthetica (MP).
  Interventions: Device: Sham High-Intensity Laser Therapy (Sham HILT)

INTERVENTIONS:
Device: High-Intensity Laser Therapy (HILT) — Participants will undergo HILT treatment using a diode laser device (wavelength: 1064 nm; power: 12 W; peak power: 50 W; energy density: 600 J/cm²; spot size: 1 cm²; pulse duration: 200 μs; pulse frequency: 10 Hz) applied in continuous mode. The laser probe will make contact with the skin over the LFCN entrapment site at three specific points: (a) the inguinal ligament, (b) the point of maximum tenderness along the nerve pathway, and (c) the mid-point between the ASIS and the lateral border of the patella. Each point will be treated for 1 minute and 40 seconds, totaling a 5-minute session. Participants will undergo 12 sessions in total, with three sessions per week for four weeks.
  Other Names: High power laser therapy
  Arms: High-Intensity Laser Therapy (HILT) Group
Device: Sham High-Intensity Laser Therapy (Sham HILT) — Participants will undergo sham HILT treatment using an identical laser device with no active laser output, following the same treatment protocol as the HILT group. The laser probe will make contact with the skin over the LFCN entrapment site at the same three specific points as the HILT group. Each point will be treated for 1 minute and 40 seconds, totaling a 5-minute session. Participants will undergo 12 sessions in total, with three sessions per week for four weeks.
  Arms: Sham High-Intensity Laser Therapy (Sham HILT) Group

SUMMARY:
This randomized controlled trial aims to investigate the efficacy of High-Intensity Laser Therapy (HILT) in the management of Meralgia Paresthetica (MP), a peripheral neuropathy causing pain, numbness, and tingling in the thigh region. Participants with MP will be randomly allocated to either the HILT or sham HILT (control) group. The study will evaluate the effects of HILT on pain intensity, functional outcomes, and quality of life. Findings from this trial will provide insights into the potential benefits of HILT as a non-invasive and safe treatment option for patients with MP.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Meralgia Paresthetica, confirmed by a neurologist or a specialist in neuromuscular disorders, based on clinical signs and symptoms, and supported by nerve conduction studies.
* Presence of pain, numbness, or tingling in the anterolateral thigh for at least three months.
* Aged between 35 and 55 years.
* Willing and able to provide informed consent.
* Able to comply with the study protocol and attend all treatment sessions and follow-up assessments.

Exclusion Criteria:

* Previous surgical treatment for Meralgia Paresthetica.
* Concomitant lower back or hip pain due to other causes, such as lumbar radiculopathy, hip joint pathology, or trochanteric bursitis.
* Presence of other neuromuscular or nerve compression disorders such as diabetic neuropathy
* Significant trauma or surgery to the affected thigh or lumbar spine within the past six months.
* Pregnancy or planning to become pregnant during the study period.
* Known contraindications to High-Intensity Laser Therapy, such as active skin infection, malignancy, or photosensitivity disorders.
* Current use of anticoagulant medications or immunosuppressive therapy.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-09-08 (Actual); Study Completion 2024-09-08 (Actual)

PRIMARY OUTCOMES:
Changes in Pain Intensity | Changes measured at Baseline, immediately post-treatment (4 weeks), and at 1- and 3-month follow-ups
  The secondary outcome measure is the change in pain intensity, assessed using the Numeric Pain Rating Scale (NPRS), a self-reported scale ranging from 0 (no pain) to 10 (worst pain imaginable). A reduction in NPRS scores indicates a decrease in pain intensity.

SECONDARY OUTCOMES:
Changes in Lateral Femoral Cutaneous Nerve Distal Latency | Changes measured at Baseline, immediately post-treatment (4 weeks), and at 1- and 3-month follow-ups
  the change in distal latency of the lateral femoral cutaneous nerve (LFCN), assessed using nerve conduction studies. The distal latency represents the time it takes for an electrical impulse to travel along the nerve to the recording electrode. Reduced distal latency indicates improved nerve conduction and function.
Changes in Functional Outcomes | Changes measured at Baseline, immediately post-treatment (4 weeks), and at 1- and 3-month follow-ups
  The secondary outcome measure is the change in functional outcomes, assessed using the Roland-Morris Disability Questionnaire (RMDQ), a self-reported questionnaire measuring the level of disability due to lower back and leg pain. Lower RMDQ scores indicate better functional outcomes and less disability.
Changes in Quality of Life | Changes measured at Baseline, immediately post-treatment (4 weeks), and at 1- and 3-month follow-ups
  The secondary outcome measure is the change in quality of life, assessed using the Short Form-36 Health Survey (SF-36), a self-reported questionnaire evaluating overall health and well-being across eight domains. Higher SF-36 scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed M ElMeligie, Ph.d, Principal Investigator — Cairo University
Locations (1):
- Outpatient clinic of faculty of physical therapy, Ahram Canadian University, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The researchers of this study are committed to promoting open science and collaboration among researchers. As part of this commitment, we will share de-identified individual participant data (IPD) with other qualified researchers, upon request and in accordance with applicable regulations and ethical guidelines. The dataset will not contain any personally identifiable information or sensitive data that could compromise the privacy and confidentiality of study participants.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified IPD will be available for sharing with other researchers starting six months after the publication of the primary study results and will remain accessible for a period of five years.
Access Criteria: Researchers interested in accessing the IPD must submit a written request to the principal investigator, detailing the information required.
  Upon approval of a request, the researchers will be required to sign a data sharing agreement that outlines the terms and conditions of IPD access, including provisions on data use, confidentiality, security, and reporting of research results.
  via email mohamed.elmeligie@acu.edu.eg